CLINICAL TRIAL: NCT01424293
Title: The Use of Fluorescent Imaging to Evaluate Bowel Anastomotic Perfusion
Brief Title: Fluorescent Evaluation of Colorectal Anastamoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Danny A Sherwinter, Attending Physician, Surgery, Maimonides Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1004va09
Record Dates: First submitted 2010-09-29; First posted 2011-08-26 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Rectal Neoplasms; Colon Neoplasms; Diverticulitis
Keywords: Rectal Cancer; Colon Cancer; Diverticulitis; Anastamosis; colectomy; low anterior resection
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms; Diverticulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indocyanine Green (Experimental): 1ml of intravenous ICG and imaging transanally using the Spyscope system
  Interventions: Device: Indocyanine Green; Device: The SPY® Intraoperative Imaging System

INTERVENTIONS:
Device: Indocyanine Green — 1ml of intravenous ICG and imaging transanally using the Spyscope system
Device: The SPY® Intraoperative Imaging System

SUMMARY:
Bowel removal is indicated for various types of colon and rectal disease, including colon cancer, rectal cancer, diverticulitis, and inflammatory bowel disease among others.

Following removal of the diseased segment of bowel your surgeon will reconnect the two healthy ends to reconstruct a continuous bowel tube. If the bowel leaks it can become an extremely dangerous situation.

The cause of leakage has many causes and is not well understood, but appears to be at least in part due to not having enough blood going to the bowel. There is currently no way to evaluate the blood supply to the bowel.

The purpose of this study is to utilize a special camera to evaluate the blood supply of the bowel. This new system is called the Spy-scope. This system may assist surgeons in reducing the occurrence of leaks

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether systemically injected ICG, when fluorescing in response to NIR illumination, can assist with the assessment of perfusion at a bowel anastomotic site. This finding may assist surgeons to minimize the occurrence of leaks at the anastomotic site following this surgical procedure. The present study is a preliminary investigation to determine if this imaging modality will yield information regarding perfusion that is likely to be clinically relevant and so determine if a larger, multi center trial that correlates perfusion to clinical outcome is warranted. The results of the present study will also assist in the design of a larger scale study. It is expected that a successful outcome to such a trial will result in less morbidity following laparoscopic colectomy.

Laparoscopic bowel surgery is indicated for colon cancer, rectal cancer, diverticulitis, inflammatory bowel disease (including ulcerative colitis or Crohn's disease) and infarcted bowel. Prophylactic colectomy is also indicated for certain forms of polyposis to mitigate the risk of progression to colon cancer. The portion of colon resected during a colectomy is dependent upon the nature of the disease and its location and extent. Traditionally, colectomy has been performed by means of laparotomy, a standard abdominal incision. In recent years, beginning in the early 1990s, there has been increasing interest in, and utilization of, minimally invasive techniques for surgical procedures involving the colon and rectum. Laparoscopic surgery involves the introduction of surgical instruments through a number (usually 2-3) of small incisions measuring about 10-12 mm each with visual guidance being provided by means of a camera attached to an endoscope introduced through a similarly small access port. Laparoscopic techniques offer numerous benefits including a decrease in postoperative pain, some improvement in time to tolerance of food and return of bowel function, shorter hospital stay and more rapid return to normal activity.

Irrespective of the type of procedure performed (open or laparoscopic), anastomotic leakage following colorectal resection and primary anastomosis is a major clinical problem. The incidence of intraperitoneal anastomotic leaks reported in the literature may be as high as 30%. Anastomotic leaks leads to increased length of hospital stay, and may progress to abscess formation, sepsis, multi organ failure and even death.

The cause of anastomotic leakage is multifactorial with the following factors appearing to impact upon leakage; adequacy of blood flow to the anastomosis, contamination, the presence of a pelvic drain, anastomotic tension, anastomotic technique and the distance from the anal verge . The present study will investigate the first factor listed above, adequacy of blood flow to the anastomosis. At present there is no reliable and easy-to-perform modality that can be used to assess adequacy of perfusion at the anastomosis during colorectal procedures. This study will investigate the potential for the SPY scope to fill this clinical need.

The SPY® Intraoperative Imaging System is cleared for use in Canada, Japan, Europe and the US. SPY was originally developed for applications in cardiac surgery and allows cardiac surgeons to visually assess bypass graft quality in real-time while the patient is still in the operating room. Subsequently, SPY has received clearance from the FDA for use in plastic and reconstructive surgery and in solid organ transplant.

The SPY Intraoperative Imaging System was originally developed for open surgical procedures using ICG, which is an approved drug. ICG is a fluorescent compound, which can be administered intravenously or intra-arterially. The dye absorbs light in the near infrared (NIR) region at 806 nm, and emits light at a slightly longer wavelength, 830 nm. When injected intravenously, ICG rapidly and extensively binds to plasma proteins and is confined to the intravascular compartment with minimal leakage into the interstitium under normal conditions. This property makes it an ideal agent for the acquisition of high quality images of the vasculature. Intraoperative images are acquired during the first pass of a bolus of ICG through the area of interest. The SPY System has been the subject of numerous peer reviewed publications demonstrating its safety and efficacy .

SPY scope, the endoscopic version of SPY, is an endoscopic visible (VIS) NIR imaging system consisting of:

* An endoscopic light source that provides illumination for visible light imaging and NIR fluorescence excitation to the endoscope via a flexible light guide
* Rigid endoscopes optimized for illuminating the field of view and transmitting images in the visible and NIR spectrum, and
* A high definition (HD) endoscopic camera system connected to the endoscope eyepiece and acquiring high resolution visible and NIR fluorescence images The ICG (25 mg per vial) will be reconstituted according to the manufacturer's instructions using the entire contents (10 ml) of the sterile diluent supplied, yielding a 2.5 mg/ml solution of ICG or using half of the diluent supplied (5 ml) yielding a 5 mg/ml solution.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for this study must meet ALL of the following inclusion criteria:

  * Subject is willing and able to provide an informed consent
  * Subject is willing and able to comply with the study procedures
  * Subject speaks English and is able to understand the study procedures
  * A pregnancy test for women of childbearing potential prior to surgery
  * Subject is scheduled for laparoscopic low anterior resection

Exclusion Criteria:

* Candidates for this study who meet any of the following criteria at the time of the baseline visit are NOT eligible to be enrolled in this study:

  * Subject has uremia, serum creatinine >2.5 mg/dl
  * Subject has a previous history of adverse reaction or allergy to ICG, iodine, shellfish or iodine dyes
  * Subjects in whom the use of x-ray dye or ICG is contraindicated including development of adverse events when previously or presently administered
  * Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
  * Subject is a pregnant or lactating female
  * Subject is actively participating in another drug, biologic and/or device protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Sherwinter, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Indocyanine Green: 1ml of intravenous ICG and imaging transanally using the Spyscope system
  Indocyanine Green: 1ml of intravenous ICG and imaging transanally using the Spyscope system
  The SPY® Intraoperative Imaging System
Period: Overall Study
Arm/Group | Indocyanine Green
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Indocyanine Green
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.29 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Vascular Supply of the Bowel Intra-operatively and Correlate This With Postoperative Complications Identified During Their Hospital Stay at One Week and One Month Postoperatively.
Description: Intra-operative evaluation of bowel perfusion. Participants will be followed for the duration of hospital stay and then at 1 week and 1 month postoperatively to identify postoperative complications.
Time Frame: 30 days
Measure: Number; unit: Complications
Arm/Group | Indocyanine Green
Number analyzed (Participants) | 7
Complications | 0

ADVERSE EVENTS:
Arm/Group | Indocyanine Green
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No